CLINICAL TRIAL: NCT01067066
Title: A Phase I/II Open-Label Study TPI 287 in Combination With Temozolomide in Patients With Metastatic Melanoma
Brief Title: A Phase I Study of TPI 287 - Temozolomide Combination in Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase I/II study halted as Phase I, Low Response Rate
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0357; NCI-2011-00558 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Melanoma
Keywords: TPI 287; microtubule inhibitor; Temozolomide; Temodar; cytotoxic agent; unresectable Stage III; Stage IV; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — TPI-287; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPI 287 + Temodar (Experimental): Starting dose of TPI 287 90 mg/m^2 IV on Days 1, 8, 15 + Temozolomide (Temodar) PO at 85 mg/m^2 on Days 1-5.
  Interventions: Drug: TPI 287; Drug: Temodar (Temozolomide)

INTERVENTIONS:
Drug: TPI 287 — Starting dose cycle 1, 90 mg/m2 by vein (IV) on Days 1, 8, 15 (+/- 1 day)
Drug: Temodar (Temozolomide) — Starting dose cycle 1, 85 mg/m^2 by mouth (PO) daily, Day 1 to 5.
  Other Names: Temozolomide

SUMMARY:
The goal of the Phase I portion of this study is to find the highest tolerable dose of TPI 287 that can be given in combination with Temodar (temozolomide) to patients with metastatic melanoma.

The goal of the Phase II portion of this study is to learn if TPI 287, given in combination with temozolomide, can control metastatic melanoma. The safety of this combination will also be studied. NOTE: Study stopped before progressing to Phase II portion.

DETAILED DESCRIPTION:
Study Drugs:

TPI 287 is designed to block tumors from growing by preventing cancer cells from dividing.

Temozolomide is designed to kill cancer cells by causing breaks in the DNA (genetic material) of the cell.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 8 groups of 6 participants will be enrolled in the Phase I portion of the study, and up to 64 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of TPI 287 and temozolomide you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of TPI 287 and temozolomide. Each new group will receive a higher dose of TPI 287 and temozolomide than the group before it, if no intolerable side effects were seen. If any of these participants have a dose limiting toxicity, 6 additional participants will be added at the same dose. If a dose limiting toxicity occurs again, the dose level below this will be considered the maximum tolerated dose.

If any participant experiences a life threatening side effect, no additional participants will be enrolled into that dose level and no higher doses will be given. An additional 3 participants will be treated at the dose level below the one with life threatening toxicity. Once the maximum tolerated dose of the combination is found, Phase II of the study will open.

If you are enrolled in the Phase II portion, you will receive the drug combination at the highest dose that was tolerated in the Phase I portion

Central Venous Catheter (CVC):

You will have a CVC placed. A CVC is a sterile, flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Study Drug Administration:

You will receive TPI 287 by vein over 1 hour (+/- 10 minutes) on Days 1, 8, and 15 (+/- 1 day) of each 28 day study cycle. Before you receive each dose of TPI 287, you will receive dexamethasone, Benadryl (diphenhydramine), and Pepcid (famotidine) by vein to help prevent allergic reaction. You will also receive drugs to prevent nausea and vomiting. Your vital signs will be measured before and 30 minutes following the end of the infusion of TPI 287. Your vitals will be measured more often, if needed.

You will take temozolomide tablets by mouth on Days 1-5 at bedtime. You should not eat for at least 1 hour before and 1 hour after taking temozolomide.

Study Visits:

Before each cycle, your performance status will be recorded and you will have a physical exam. You will also be asked about any symptoms you may be experiencing and any drugs you are taking.

On Days 1, 8, and 14 of each cycle:

-Blood (about 1 teaspoon) will be drawn for routine tests before you receive TPI 287.

On Day 22 of each cycle:

-Blood (about 1 teaspoon) will be drawn for routine tests.

Every 8 weeks, you will have a CT scan or MRI scan to check the status of the disease. If you have brain metastasis, you will have an MRI of the brain every 4 weeks. If you do not have brain metastasis, you will have MRI of the brain every 8 weeks.

Length of Study:

You will continue taking the study drugs for as long as you are benefitting. You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

About 4 weeks after you stop taking TPI 287 in combination with Temozolomide, you have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* You will be asked about any complications or side effects you may be experiencing.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a CT scan or MRI scan to check the status of the disease.

This is an investigational study. TPI 287 is not FDA approved or commercially available. At this time, TPI 287 is being used in research only. Temozolomide is FDA approved and commercially available for primary brain cancer. The use of temozolomide in combination with TPI 287 is investigational.

Up to 106 patients will take part in this study. All patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven melanoma with metastasis that is unresectable Stage III or Stage IV. This will include bulky stage III and M1-3. Patients with melanoma with documented metastases to the brain are eligible.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression and should have at least one indicator lesion, that can be measured in one dimension as >/=20mm with conventional techniques (CT, MRI, X-ray) or >/=10mm with spiral CT scan.
3. Patients may have had up to two prior cytotoxic chemotherapy regimens for their disease (immunological or targeted therapy e.g. vaccine, IL-2, B-RAF inhibitors, will not be considered prior cytotoxic chemotherapy). Patient should not have been treated with Docetaxel, Paclitaxel or other taxanes.
4. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
5. Patients must have a Eastern Cooperative Oncology Group status of </=2.
6. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
7. Patients must have adequate bone marrow function (ANC >/= 1,500/mm3 and platelet count of >/= 100,000/mm3), adequate liver function (SGPT and serum glutamate oxaloacetate transaminase (SGOT) </= 2.5 times normal, bilirubin </= 2 mg/dl), and adequate renal function (BUN and creatinine </=1.5 times institutional normal) prior to starting therapy.
8. TPI 287 may interfere with coumadin dosing and patients who are taking this combination will require monitoring of their PT, PTT and international normalized ratio (INR).
9. Females of childbearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods (abstinence, intrauterine device, oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.
10. Patient should be 15 years of age or older

Exclusion Criteria:

1. Patients with brain metastases must not be taking primidone, carbamazepine, phenobarbital or phenytoin anticonvulsants (Enzyme-Inducing Anti-Epileptic Drugs). Patients changing from these anticonvulsants to others that are allowed must be off the drugs listed above for at least 1 week.
2. Patients with any neuropathy.
3. Patients with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, history of myocardial infarction within the previous six months, or serious uncontrolled cardiac arrhythmia.
4. Because of the concerns of potentially harmful interactions of TPI 287and other medications taken by patients who are HIV positive or have AIDS related diseases, patients who are HIV positive are not be eligible for entry into this study. Only patients with suspected HIV will be tested and if positive, will be ineligible.
5. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) are ineligible for Phase II part of the study unless in complete remission and off of all therapy for that disease for a minimum of 3 years. However, during Phase I part of the study, a patient with second malignancy is eligible if that malignancy has not recurred after appropriate therapy.
6. Patients with: a) active infection, b) disease that will obscure toxicity or dangerously alter drug metabolism, c) serious intercurrent medical illness, d) prior documented recurrence with temozolomide
7. Females who are pregnant or breastfeeding.
8. Patients younger than 15 years of age
9. Patients with prior therapy with paclitaxel or other taxanes.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02-03 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of TPI 287 in Combination with Temodar | 28 day study cycle
  MTD is highest dose level in which 6 patients treated with at most 1 experiencing dose limiting toxicity (DLT).
  Maximum Tolerated Dose (MTD), measured by clinical and laboratory adverse events.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Response rate provided along with a 95% credible interval. Logistic regression models used to assess the association between progression-free survival at 6 months and covariates of interest. Additionally, Cox proportional hazards regression models will be fit to model the association between progression-free survival and the same covariates. Simon's minimax two-stage design used to evaluate the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org